## A Randomized Controlled Study to Explore the Clinical Effect of Intermittent Oro-esophageal Tube Feeding vs. Nasogastric Tube Feeding on Cerebral Small Vessel Disease Patients with Dysphagia

Plan number

Version V1.0

Date 2022.12.10

Research unit Department of Rehabilitation Medicine,

The First Affiliated Hospital of Zhengzhou

University

Main Researchers Zengxi

Research responsible unit The First Affiliated Hospital of Zhengzhou

University

Applicant Department of Rehabilitation Medicine,

The First Affiliated Hospital of Zhengzhou

University

The measurement data with normal distribution obtained in this study were represented in the form of  $(x \pm s)$ , while those with skewed distribution were expressed as medians and quartiles (m, q). A t-test or Mann-Whitney U test were recruited accordingly to analyze the difference. Categorical data and grade data were expressed as number of cases and percentage (n, %) and Chi-square tests or Mann-Whitney U test were performed accordingly. Besides, we conducted Fisher's exact tests instead of Chi-square tests to categorical data when there was at least one minimum theoretical frequency T <1. SPSS 21.0 statistical was used for analysis and a p-value of less than 0.05 was regarded as the existence of statistical significance.